CLINICAL TRIAL: NCT02877420
Title: Impact of a Simulation-based Training Curriculum of Non-technical Skills on Colonoscopy Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Samir Grover, MD, MEd, FRCPC, Unity Health Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 15-164c
Record Dates: First submitted 2016-07-28; First posted 2016-08-24 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Endoscopy Simulation
Keywords: Endoscopy; Simulation Training; Non-technical Skills

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-Technical Skills Training Curriculum (Experimental): This group will receive 4 hours of small-group and hands-on sessions and 1 hour of didactic NTS sessions. Participants will watch a video that demonstrates ideal endoscopic performance. They will use the E-NTS Checklist during the integrated scenario training. This checklist targets NTS. The group will be given 7 hours of expert-assisted instruction on the low-fidelity simulator (1 hour) and the high-fidelity VR simulator (6 hours). Six modules of increasing difficulty in colonoscopy and polypectomy will be taught with feedback from an expert endoscopist who will demonstrate techniques, answer questions and provide individualized performance feedback with a focus on NTS. The last three hours on the high fidelity simulator will be an integrated scenario (IG) featuring standardized patient (SP) and standardized nurse (SN). Feedback will be given after each IG by the instructor, SP and SN. Participants can view the E-NTS Checklist before and after each case.
  Interventions: Other: Non-Technical Skills Training Curriculum
- Conventional Simulation Training Group (Active Comparator): This group will receive 4 hours of small-group and hands-on sessions on colonoscopy theory from an expert endoscopist. The core curriculum is designed on the basis of the American Society for Gastrointestinal Endoscopy colonoscopy curriculum and an endoscopic training textbook. This curriculum has been shown to be effective when compared to self-regulated learning on the simulator. The sessions will be interlaced with eight hours of expert-assisted instruction on both the low-fidelity simulator (1 hour) and on the high-fidelity VR simulator (7 hours). Six modules of increasing difficulty in colonoscopy and polypectomy will be taught with feedback from an expert endoscopist. The expert will demonstrate techniques, answer questions and provide feedback on global performance. Feedback, in the form of performance metrics, will be provided by the simulator upon completion/failure of each module.
  Interventions: Other: Conventional Simulation Training Group

INTERVENTIONS:
Other: Non-Technical Skills Training Curriculum
  Arms: Non-Technical Skills Training Curriculum
Other: Conventional Simulation Training Group
  Arms: Conventional Simulation Training Group

SUMMARY:
The investigators aim to test a curriculum of non-technical skills (NTS) training for simulation-based training of colonoscopy. There is no known literature to date on the optimal approach on how to teach NTS in endoscopy. The objectives are to evaluate a simulation-based curriculum to teach NTS, to explore the relationship between NTS and other domains of competency, and understand how NTS are acquired in endoscopic training.

DETAILED DESCRIPTION:
This study will employ a randomized controlled two-arm design. All testing and training will take place at St. Michael's Hospital (30 Bond Street, Toronto, Ontario). During the study participants will be performing simulated lower endoscopic procedures on a virtual reality (VR) endoscopy simulator.

Description of Simulation Devices used

Low-Fidelity Simulator (Bench Top Model): The low-fidelity simulator is a validated bench-top endoscopy simulator that helps develop general endoscopic skills. The simulator is comprised of a series of vertical wooden barriers with numbered targets (holes) conforming to 27 different sequences of varying complexity. An Olympus paediatric videocolonoscope is used to navigate the defined sequences as quickly and accurately as possible, with visual output being displayed on a video monitor.

High-Fidelity Simulator: Virtual Reality Model: The high-fidelity simulator to be used for testing and training is the EndoVR® virtual reality (VR) endoscopy simulator. It models navigation through a colon, using a specialized endoscope that is inserted into a computer-based module with a screen showing the colonic lumen of a virtual patient. It provides both visual and haptic feedback related to the procedure. The VR simulator has a number of standardized case-based scenarios of varying complexity for colonoscopy.

Details of experimental design

Baseline questionnaire: A written questionnaire will be administered to all participants at the start of the project to collect demographic and background information including: age, sex, level of training, previous endoscopy experience and nature of experience (if applicable), and video game experience, which may correlate with baseline endoscopic skill.

Pre-test: All participants will then take part in a pre-test designed to assess their baseline (1) knowledge of colonoscopy; (2) technical skills; and (3) non-technical skills. No feedback will be provided at any point during the pre-test. The pre-test will consist of the following:

Knowledge Test: A 30 minute (20 questions) multiple-choice question test designed to assess participants' theoretical knowledge of colonoscopy, including indications, sedation, safety, findings, pathology and follow-up.

VR Simulation Test: Participants baseline endoscopic technical proficiency will be will be assessed through the completion of a colonoscopy procedure on the VR simulator. This scenario simulates a screening colonoscopy, without the need for any type of intervention such as biopsy. The procedure will be timed so that participants do not take longer than 30 minutes to complete the procedure. An expert rater will be present to assess performance, but will not provide assistance. All participants will be videotaped in order to obtain performance measures such that their faces are not captured to ensure anonymity. Prior to starting the procedure, participants will complete a questionnaire to measure their self-efficacy.

VR Simulation Based "Integrated Scenario" Test: Following the simulator-only test, participants will complete an Integrated Scenario format test to assess their baseline endoscopic non-technical proficiency. This test was modeled after another test during which participants perform a colonoscopy procedure on the VR simulator while interacting with an endoscopic nurse and a standardized patient (SP) portraying a patient. The simulated procedure will mimic the setup of an endoscopic suite, as the VR simulator will be positioned next to a patient bed. A standardized patient, who will receive instructions regarding their medical role, will act out a scenario on colon cancer screening. Trainees will be expected to explain the colonoscopy procedure, its benefits and risks, and obtain procedural consent. The trainee will then carry out the procedure on the VR simulator while responding to the patient and interacting with the standardized nurse (SN) as appropriate. The SP will act out cues from the VR simulator if the simulator signals that the procedure has exceeded its threshold for discomfort. The performance of all participants will be videotaped (in a manner that their faces are not captured to ensure anonymity) in order to obtain performance measures. Participants will be given a maximum of 45 minutes to complete the procedure. Prior to starting the procedure, participants will complete a questionnaire to measure their self-efficacy.

Training interventions: Subsequently participants will be randomized, using an online randomization algorithm, to one of two groups (following a 1:1 allocation distribution)

Sample size calculation: A power analysis was computed using G*Power version 3.1.9. Using a previous study that evaluated an NTS training curriculum in surgery as assessed by the Non-Technical Skills for Surgeons (NOTSS) and OSANTS forms, we conducted the analysis using the relevant effect size. Based on an effect size of 0.65 (effect size f), an alpha of 0.05 (two-tailed), a beta of 0.20, 2 groups, and 3 measurements, 16 participants are required to achieve a power of greater than 0.80 using repeated measures ANOVA (between-factors). Furthermore, a previous study comparing a curriculum in endoscopic simulation found that a minimum of 15 participants per group was sufficient to detect a significant difference. To accommodate for a projected 20% dropout and/or non-response that may occur, we therefore plan to recruit a total of 36 participants.

Statistical analysis: Statistical analyses will be performed using Statistical Package for the Social Sciences (SPSS) version 20. All statistical tests will be considered significant at p < 0.05. Baseline Questionnaire: Patient demographics and baseline variables will be compared between the two groups using Analysis of Variance (ANOVA) and chi-square tests for continuous and categorical variables respectively. (b)Clinical Performance (Technical and Non-Technical): Clinical performance during the live colonoscopies for each group will be determined by comparing the scores from the DOPS, GiECAT, NAPCOMS, and Modified-OSANTS. Specifically, a mixed factor 2 (NTS curriculum vs. TS curriculum) x 2 (procedure 1 vs. procedure 2) ANOVA will be used to determine whether there is a difference based on the rating scales. Tukey's honest significant difference (HSD) test will be used as a post-hoc analysis to determine any significant differences.

Technical Performance: Technical performance on the simulator for each group will be determined by comparing the scores from the DOPS, GiECAT, and GAGES. Specifically, a mixed factor 2 (NTS curriculum vs. TS curriculum) x 3 (pretest, posttest, retention test) ANOVA will be used to determine whether there is a difference based on the rating scales. Tukey HSD test will be used as a post-hoc analysis to determine any significant differences.

Non-Technical Performance: Non-technical performance on the simulator for each group will be determined by comparing the scores from the GiECAT and modified OSANTS. Specifically, a mixed factor 2 (NTS curriculum vs. TS curriculum) x 3 (pretest, posttest, retention test) ANOVA will be used to determine whether there is a difference based on the rating scales. Tukey HSD test will be used as a post-hoc analysis to determine any significant differences.

ELIGIBILITY:
Inclusion Criteria:

* Novice endoscopists from general surgery, gastroenterology, or pediatrics gastroenterology residency programs at the University of Toronto

Exclusion Criteria:

* If participants have performed more than 25 endoscopies

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Difference in performance between two groups in clinical colonoscopy | During clinical colonoscopy 4-6 weeks after NTS training curriculum
  Each videotaped clinical colonoscopy will be independently assessed by two experienced endoscopists using the Joint Advisory Group for GI Endoscopy Direct Observation of Procedural Skills (JAG/DOPS). The raters will be blinded to the group assignment. Training on how to use the tool will be provided for raters by the investigators of the study.

SECONDARY OUTCOMES:
Differences in procedural knowledge | One day
  Assessed through multiple choice question tests
Technical performance on a VR simulated colonoscopy - JAG/DOPS | 4-6 weeks
  Assessed through a Joint Advisory Group for GI Endoscopy Direct Observation of Procedural Skills (JAG/DOPS).
Technical performance on a VR simulated colonoscopy - GiECAT | 4-6 weeks
  Assessed through the Gastrointestinal Endoscopy Competency Assessment Tool for Pediatric Colonoscopy (GiECAT).
Patient comfort during clinical colonoscopies | 4-6 weeks
  Assessed through Nurse-Assessed Patient Comfort Score (NAPCOMS).
Non-technical performance on clinical colonoscopies | 4-6 weeks
  Assessed through the Modified Objective Structured Assessment of Nontechnical Skills (MOSANTS)
Clinical performance on clinical colonoscopies - GiECAT | 4-6 weeks
  Assessed through GiECAT
Participant self-efficacy | 1 day
  Assessed through an adapted scale based on the General Self-Efficacy Scale.
Practice case length on simulator | 1 day
  Assessed through a time measurement of the length of the case. Experienced endoscopists will assess participants' colonoscopy-specific skills, technical skills and non-technical skills during the pre-training, immediate and delayed post-training simulation-based assessments

CONTACTS AND LOCATIONS:
Overall Officials: Samir C Grover, MD, MEd, Principal Investigator — Unity Health Toronto
Locations (1):
- St.Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arriaga AF, Bader AM, Wong JM, Lipsitz SR, Berry WR, Ziewacz JE, Hepner DL, Boorman DJ, Pozner CN, Smink DS, Gawande AA. Simulation-based trial of surgical-crisis checklists. N Engl J Med. 2013 Jan 17;368(3):246-53. doi: 10.1056/NEJMsa1204720. PMID 23323901
- [Background] Bandura A. Self-efficacy: toward a unifying theory of behavioral change. Psychol Rev. 1977 Mar;84(2):191-215. doi: 10.1037//0033-295x.84.2.191. No abstract available. PMID 847061
- [Background] Barton JR, Corbett S, van der Vleuten CP; English Bowel Cancer Screening Programme; UK Joint Advisory Group for Gastrointestinal Endoscopy. The validity and reliability of a Direct Observation of Procedural Skills assessment tool: assessing colonoscopic skills of senior endoscopists. Gastrointest Endosc. 2012 Mar;75(3):591-7. doi: 10.1016/j.gie.2011.09.053. Epub 2012 Jan 9. PMID 22227035
- [Background] Brydges R, Carnahan H, Rose D, Rose L, Dubrowski A. Coordinating progressive levels of simulation fidelity to maximize educational benefit. Acad Med. 2010 May;85(5):806-12. doi: 10.1097/ACM.0b013e3181d7aabd. PMID 20520031
- [Background] Cook TM, Woodall N, Harper J, Benger J; Fourth National Audit Project. Major complications of airway management in the UK: results of the Fourth National Audit Project of the Royal College of Anaesthetists and the Difficult Airway Society. Part 2: intensive care and emergency departments. Br J Anaesth. 2011 May;106(5):632-42. doi: 10.1093/bja/aer059. Epub 2011 Mar 29. PMID 21447489
- [Background] Dedy NJ, Bonrath EM, Ahmed N, Grantcharov TP. Structured Training to Improve Nontechnical Performance of Junior Surgical Residents in the Operating Room: A Randomized Controlled Trial. Ann Surg. 2016 Jan;263(1):43-9. doi: 10.1097/SLA.0000000000001186. PMID 25775073
- [Background] Dedy NJ, Szasz P, Louridas M, Bonrath EM, Husslein H, Grantcharov TP. Objective structured assessment of nontechnical skills: Reliability of a global rating scale for the in-training assessment in the operating room. Surgery. 2015 Jun;157(6):1002-13. doi: 10.1016/j.surg.2014.12.023. Epub 2015 Feb 20. PMID 25704419
- [Background] Faul F, Erdfelder E, Buchner A, Lang AG. Statistical power analyses using G*Power 3.1: tests for correlation and regression analyses. Behav Res Methods. 2009 Nov;41(4):1149-60. doi: 10.3758/BRM.41.4.1149. PMID 19897823
- [Background] Flin R, Patey R, Glavin R, Maran N. Anaesthetists' non-technical skills. Br J Anaesth. 2010 Jul;105(1):38-44. doi: 10.1093/bja/aeq134. Epub 2010 Jun 3. PMID 20522911
- [Background] Flin R, Yule S, Paterson-Brown S, Maran N, Rowley D, Youngson G. Teaching surgeons about non-technical skills. Surgeon. 2007 Apr;5(2):86-9. doi: 10.1016/s1479-666x(07)80059-x. PMID 17450689
- [Background] Gordon M, Darbyshire D, Baker P. Non-technical skills training to enhance patient safety: a systematic review. Med Educ. 2012 Nov;46(11):1042-54. doi: 10.1111/j.1365-2923.2012.04343.x. PMID 23078681
- [Background] Grover SC, Garg A, Scaffidi MA, Yu JJ, Plener IS, Yong E, Cino M, Grantcharov TP, Walsh CM. Impact of a simulation training curriculum on technical and nontechnical skills in colonoscopy: a randomized trial. Gastrointest Endosc. 2015 Dec;82(6):1072-9. doi: 10.1016/j.gie.2015.04.008. Epub 2015 May 23. PMID 26007221
- [Background] Guadagnoli MA, Lee TD. Challenge point: a framework for conceptualizing the effects of various practice conditions in motor learning. J Mot Behav. 2004 Jun;36(2):212-24. doi: 10.3200/JMBR.36.2.212-224. PMID 15130871
- [Background] Guadagnoli M, Morin MP, Dubrowski A. The application of the challenge point framework in medical education. Med Educ. 2012 May;46(5):447-53. doi: 10.1111/j.1365-2923.2011.04210.x. PMID 22515752
- [Background] Hales B, Terblanche M, Fowler R, Sibbald W. Development of medical checklists for improved quality of patient care. Int J Qual Health Care. 2008 Feb;20(1):22-30. doi: 10.1093/intqhc/mzm062. Epub 2007 Dec 11. PMID 18073269
- [Background] Hatala R, Cook DA, Zendejas B, Hamstra SJ, Brydges R. Feedback for simulation-based procedural skills training: a meta-analysis and critical narrative synthesis. Adv Health Sci Educ Theory Pract. 2014 May;19(2):251-72. doi: 10.1007/s10459-013-9462-8. Epub 2013 May 28. PMID 23712700
- [Background] Hoch JS, Rockx MA, Krahn AD. Using the net benefit regression framework to construct cost-effectiveness acceptability curves: an example using data from a trial of external loop recorders versus Holter monitoring for ambulatory monitoring of "community acquired" syncope. BMC Health Serv Res. 2006 Jun 6;6:68. doi: 10.1186/1472-6963-6-68. PMID 16756680
- [Background] Hull L, Arora S, Aggarwal R, Darzi A, Vincent C, Sevdalis N. The impact of nontechnical skills on technical performance in surgery: a systematic review. J Am Coll Surg. 2012 Feb;214(2):214-30. doi: 10.1016/j.jamcollsurg.2011.10.016. Epub 2011 Dec 24. PMID 22200377
- [Background] Kemper PF, van Noord I, de Bruijne M, Knol DL, Wagner C, van Dyck C. Development and reliability of the explicit professional oral communication observation tool to quantify the use of non-technical skills in healthcare. BMJ Qual Saf. 2013 Jul;22(7):586-95. doi: 10.1136/bmjqs-2012-001451. Epub 2013 Feb 14. PMID 23412933
- [Background] Kneebone R, Nestel D, Yadollahi F, Brown R, Nolan C, Durack J, Brenton H, Moulton C, Archer J, Darzi A. Assessing procedural skills in context: Exploring the feasibility of an Integrated Procedural Performance Instrument (IPPI). Med Educ. 2006 Nov;40(11):1105-14. doi: 10.1111/j.1365-2929.2006.02612.x. PMID 17054620
- [Background] Mann KV. Theoretical perspectives in medical education: past experience and future possibilities. Med Educ. 2011 Jan;45(1):60-8. doi: 10.1111/j.1365-2923.2010.03757.x. PMID 21155869
- [Background] Matharoo M, Haycock A, Sevdalis N, Thomas-Gibson S. Endoscopic non-technical skills team training: the next step in quality assurance of endoscopy training. World J Gastroenterol. 2014 Dec 14;20(46):17507-15. doi: 10.3748/wjg.v20.i46.17507. PMID 25516665
- [Background] Matharoo M, Sevdalis N, Thillai M, Bouri S, Marjot T, Haycock A, Thomas-Gibson S. The endoscopy safety checklist: A longitudinal study of factors affecting compliance in a tertiary referral centre within the United Kingdom. BMJ Qual Improv Rep. 2015 Feb 11;4(1):u206344.w2567. doi: 10.1136/bmjquality.u206344.w2567. eCollection 2015. PMID 26734331
- [Background] Mishra A, Catchpole K, McCulloch P. The Oxford NOTECHS System: reliability and validity of a tool for measuring teamwork behaviour in the operating theatre. Qual Saf Health Care. 2009 Apr;18(2):104-8. doi: 10.1136/qshc.2007.024760. PMID 19342523
- [Background] Pena G, Altree M, Field J, Thomas MJ, Hewett P, Babidge W, Maddern GJ. Surgeons' and trainees' perceived self-efficacy in operating theatre non-technical skills. Br J Surg. 2015 May;102(6):708-15. doi: 10.1002/bjs.9787. Epub 2015 Mar 19. PMID 25790065
- [Background] Reader T, Flin R, Lauche K, Cuthbertson BH. Non-technical skills in the intensive care unit. Br J Anaesth. 2006 May;96(5):551-9. doi: 10.1093/bja/ael067. Epub 2006 Mar 27. PMID 16567346
- [Background] Rostom A, Ross ED, Dube C, Rutter MD, Lee T, Valori R, Bridges RJ, Pontifex D, Webbink V, Rees C, Brown C, Whetter DH, Kelsey SG, Hilsden RJ. Development and validation of a nurse-assessed patient comfort score for colonoscopy. Gastrointest Endosc. 2013 Feb;77(2):255-61. doi: 10.1016/j.gie.2012.10.003. PMID 23317691
- [Background] Savoldelli GL, Naik VN, Park J, Joo HS, Chow R, Hamstra SJ. Value of debriefing during simulated crisis management: oral versus video-assisted oral feedback. Anesthesiology. 2006 Aug;105(2):279-85. doi: 10.1097/00000542-200608000-00010. PMID 16871061
- [Background] Undre S, Healey AN, Darzi A, Vincent CA. Observational assessment of surgical teamwork: a feasibility study. World J Surg. 2006 Oct;30(10):1774-83. doi: 10.1007/s00268-005-0488-9. PMID 16983480
- [Background] van Dongen KW, Verleisdonk EJ, Schijven MP, Broeders IA. Will the Playstation generation become better endoscopic surgeons? Surg Endosc. 2011 Jul;25(7):2275-80. doi: 10.1007/s00464-010-1548-2. Epub 2011 Mar 17. PMID 21416186
- [Background] Walsh CM, Ling SC, Khanna N, Grover SC, Yu JJ, Cooper MA, Yong E, Nguyen GC, May G, Walters TD, Reznick R, Rabeneck L, Carnahan H. Gastrointestinal Endoscopy Competency Assessment Tool: reliability and validity evidence. Gastrointest Endosc. 2015;81(6):1417-1424.e2. doi: 10.1016/j.gie.2014.11.030. Epub 2015 Mar 7. PMID 25753836
- [Background] Walsh CM, Ling SC, Walters TD, Mamula P, Lightdale JR, Carnahan H. Development of the gastrointestinal endoscopy competency assessment tool for pediatric colonoscopy (GiECAT KIDS). J Pediatr Gastroenterol Nutr. 2014 Oct;59(4):480-6. doi: 10.1097/MPG.0000000000000358. PMID 24590220
- [Background] Walsh CM, Sherlock ME, Ling SC, Carnahan H. Virtual reality simulation training for health professions trainees in gastrointestinal endoscopy. Cochrane Database Syst Rev. 2012 Jun 13;(6):CD008237. doi: 10.1002/14651858.CD008237.pub2. PMID 22696375
- [Background] Yule S, Flin R, Paterson-Brown S, Maran N. Non-technical skills for surgeons in the operating room: a review of the literature. Surgery. 2006 Feb;139(2):140-9. doi: 10.1016/j.surg.2005.06.017. PMID 16455321
- [Derived] Khan R, Scaffidi MA, Walsh CM, Lin P, Al-Mazroui A, Chana B, Kalaichandran R, Lee W, Grantcharov TP, Grover SC. Simulation-Based Training of Non-Technical Skills in Colonoscopy: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2017 Aug 4;6(8):e153. doi: 10.2196/resprot.7690. PMID 28778849